CLINICAL TRIAL: NCT05073094
Title: Myocardial Protection With Esmolol in Patients With Hypertrophic Obstructive Cardiomyopathy Undergoing Surgery Under Cardiopulmonary Bypass
Brief Title: Esmolol for Myocardial Protection in Hypertrophic Obstructive Cardiomyopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BETABLOCK-21
Record Dates: First submitted 2021-05-19; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — esmolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esmolol (Experimental): 1 mg/kg (max. 100 mg) as a bolus before aortic cross-clamping and 2 mg/kg (max. 200 mg) in the cardioplegia solution
  Interventions: Drug: Esmolol
- Placebo (Placebo Comparator): Equivalent volume of saline as a bolus before aortic cross-clamping and in the cardioplegic solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esmolol — Esmolol injected intravenously and added to cardioplegia solution
  Arms: Esmolol
Drug: Placebo — Equivalent volume of placebo (saline) as a bolus before aortic cross-clamping and in the cardioplegic solution
  Arms: Placebo

SUMMARY:
Perioperative blockage of beta-adrenoreceptors is widely used in cardiac and non-cardiac surgery to reduce the rate of cardiovascular complications. Several randomized-controlled studies and meta-analysis showed that esmolol reduces the incidence of myocardial ischemia and arrhythmias in cardiac surgery as well as enhances postoperative cardiac performance. No studies assessed the influence of esmolol in patients with hypertrophic obstructive cardiomyopathy undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Signed informed consent
* Patient with hypertrophic obstructive cardiomyopathy undergoing surgery under cardiopulmonary bypass

Exclusion Criteria:

* History of adverse effects on esmolol
* Urgent/emergent surgery
* Administration of esmolol in 30 days before randomization
* Participation in other randomized trial during same hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Peak concentration of Troponin I | From the randomization to the postoperative day 3 (POD 3)

SECONDARY OUTCOMES:
The need for (yes/no) inotropic agents | through study completion, an average of 4 weeks
  Number of patients requiring inotropic support
The need for (yes/no) defibrillation | through study completion, an average of 4 weeks
  Number of patients requiring defibrlillation after removal of aortic cross clamp
The incidence of new-onset moderate and severe arrhythmias of cardiac arrest | through study completion, an average of 4 weeks
  Number of patients with arrhythmias
Left ventricular ejection fraction | through study completion, an average of 4 weeks
Peak serum creatinine concentration | through study completion, an average of 4 weeks
The incidence of acute kidney injury | through study completion, an average of 4 weeks
Duration of mechanical ventilation | through study completion, an average of 4 weeks
Duration of ICU stay | through study completion, an average of 4 weeks
Duration of hospital stay | through study completion, an average of 4 weeks
30-day all-cause mortality | through study completion, an average of 4 weeks
Presence of diastolic dysfunction | through study completion, an average of 4 weeks
The dosage of inotropic agents (inotropic score) | through study completion, an average of 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- E. Meshalkin National Medical Research Center, Novosibirsk, Russia

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33451954/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27932571/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29398384/